CLINICAL TRIAL: NCT02749721
Title: Relationship Among Changes in Brain Network Activation, Changes in Core Depressive and Cognitive Symptoms and Safety and Tolerability in Adults With Major Depressive Disorder Treated With Open-Label, Flexible-Dose Vortioxetine
Brief Title: The Relationship Among Changes in Brain Network Activation in Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry); ElMindA Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IISR-2014-100702a; NCT02559947 (obsolete NCT alias)
Record Dates: First submitted 2016-04-14; First posted 2016-04-25 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
Keywords: depression; brain network activation; vortioxetine
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Other - vortioxetine (Other): Open-label vortioxetine
  Interventions: Drug: vortioxetine

INTERVENTIONS:
Drug: vortioxetine — Open-label vortioxetine

SUMMARY:
The purpose of this study is to explore patterns of Brain Network Activation (BNA) changes from baseline to endpoint on 1) efficacy of core symptoms of Major Depressive Disorder (MDD) and 2) improvement of cognitive dysfunction with acute treatment with flexible dose vortioxetine in adult outpatients with MDD and subjective complaints of cognitive dysfunction.

DETAILED DESCRIPTION:
Vortioxetine is a novel antidepressant with hypothetical multimodal mechanism of action. It is thought to work through a combination of multiple pharmacological modes of action: 5-HT (hydroxytryptamine, or serotonin) reuptake inhibition, 5-HT3 (hydroxytryptamine, or serotonin) and 5-HT7 (hydroxytryptamine, or serotonin) receptor antagonism, 5-HT1A (hydroxytryptamine, or serotonin) receptor agonism, and 5-HT1B (hydroxytryptamine, or serotonin) receptor partial agonism. In vivo nonclinical studies have demonstrated that vortioxetine enhances levels of the neurotransmitters 5-HT (hydroxytryptamine, or serotonin), norepinephrine (NE), dopamine (DA), acetylcholine and histamine in specific areas of the brain. These affinities are all considered to be of clinical relevance and involved in the mechanism of action at therapeutic doses.

Vortioxetine has been shown to improve core depressive symptoms and improve cognitive function in adult outpatients with MDD and subjective complaints of cognitive function. This pilot study is intended to evaluate the extent to which BNA technology can provide clinically valuable information and provide information toward designing a subsequent confirmatory study that will further elucidate the effect of vortioxetine on MDD and cognitive function in this population. This exploratory study will ascertain the acute changes in core depression symptoms, cognitive function, tolerability, and safety using flexible-dose vortioxetine in adult outpatients with MDD with subjective complaints of cognitive functioning, as measured by BNA changes and standard outcome measures for depression and cognition.

The study consists of 8 weeks of open-label treatment for MDD with response to treatment measured by standard research depression scales and BNA electroencephalogram (EEG) readings taken at certain points during the trial. An important aim in this study is to explore what correlations may exist between changes in measured brainwave patterns and reported change in depressive symptoms

ELIGIBILITY:
Inclusion Criteria:

* The subject has single episode or recurrent MDD (acute onset of recurrence of recurrent MDD with poor inter-episode recovery) (inter-episode periods cannot meet full MDD criteria) as the primary diagnosis according to DSM-IV-TR criteria. The current major depressive episode (MDE) will be confirmed using the Mini International Neuropsychiatric Interview (MINI V6.0.0).
* The subject has a MADRS total score ≥26.
* Subject reports subjective cognitive dysfunction (such as difficulty concentrating, slow thinking, and difficulty in learning new things or remembering things).
* The reported duration of the current MDE is at least 3 months and no longer than 24 months.
* The subject is a man or woman between 18 and 65 years old, inclusive.
* Right-handed, normal (corrected) vision, and normal hearing.

Exclusion Criteria:

* The subject has a score of ≥70 on the Digit Symbol Substitution Test (DSST) at the Baseline Visit.
* Failure to respond to or inability to tolerate an adequate trial of vortioxetine in the past.
* Exposure to an investigational compound 30 days prior to enrollment
* Exposure to any psychoactive or otherwise excluded medication within five half-lives of the baseline visit or during the study. Excluded medications include: antidepressants, anxiolytics, anticonvulsants, barbiturates, chloral hydrate, lithium, antipsychotics, benzodiazepines, hypnotics, monoamine oxidase inhibitors (MAOIs), muscle relaxers, triptans, centrally-acting antihistamines, central alpha-2 agonists, decongestants, psychostimulants, dopamine agonists, opioid pain medications, oral corticosteroids, L-methylfolate, S-adenosyl methionine (SAMe), 5-HTP (hydroxytryptophan), St. John's Wort,
* The subject has 1 or more of the following:

  * Primary psychiatric disorder other than MDD as defined in the Diagnostic and Statistical Manual of Mental Disorders 4 Text Revision (DSM-IV-TR) (as assessed by the MINI, Version 6.0.0).
  * Current or history of attention deficit hyperactivity disorder (ADHD), pervasive developmental disorder, manic or hypomanic episode, schizophrenia, or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Current diagnosis of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in sustained full remission for at least 6 months (for abuse) and 12 months (for dependence) prior to Screening.
  * Positive urine drug screen prior to Baseline.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer Disease, Parkinson Disease, multiple sclerosis, Huntington Disease, etc).
  * Any unstable medical condition as determined by the principal investigator (PI).
  * Any DSM-IV Axis II disorder that might compromise the study as determined by the PI.
* The subject has any other disorder for which the treatment takes priority over treatment of MDD or is likely to interfere with study treatment or impair treatment compliance.
* The subject has physical, cognitive, or language impairment of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
* The subject has a significant risk of suicide according to the PI's clinical judgment.
* The subject, in the opinion of the PI, poses a risk of harm to others.
* The subject has initiated formal cognitive or behavioral therapy, systemic psychotherapy within less than 6 months of study screening, or has plans to initiate such therapy during the study.
* The subject has received electroconvulsive therapy, vagus nerve stimulation, or repetitive transcranial magnetic stimulation within 12 months prior to Screening.
* The current MDE is considered by the PI to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each at the recommended dose.
* The subject is pregnant or breastfeeding, or is intending to become pregnant before, during, or within 30 days after participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Zajecka, MD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Rush University Medical Center, Skokie, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from several sources, including referrals, advertisements and following completion of another clinical trial.
Pre-assignment Details: Participants were screened over a 1-2 week period to assess inclusion/exclusion criteria (i.e., to obtain lab results, to ensure adequate washout of any prohibited concomitant medications, etc).
Groups:
- Vortioxetine: vortioxetine 5-20 mg/day
Period: Screening
Arm/Group | Vortioxetine
Started | 31
Completed | 25
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 3
Period: 8-week Open-Label Treatment Phase
Arm/Group | Vortioxetine
Started | 25
Completed | 22
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Major Depressive Disorder-single or recurrent [Number; unit: participants]
  Recurrent episode | 19
  Single episode | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery and Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item rating scale designed to assess the severity of symptoms of depression. Range is 0-60. Higher score means more severe.
Time Frame: from baseline to endpoint (up to 8 weeks)
Population: 25 subjects were included in the baseline analysis, and 22 subjects completed all visits and were included in subsequent analyses
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
score on a scale
  Baseline | 33.28 [24 to 40]
  Week 8: number analyzed (Participants) | 22
  Week 8 | 16.23 [2 to 31]
Statistical Analysis 1: Comparison: Vortioxetine; Test type: Other; p < 0.001, Paired t-test

2. Primary Outcome: Change From Baseline to Endpoint in Digital Symbol Substitution Test.
Description: Change in cognitive function defined as change from baseline to endpoint. The Digital Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making and motor skills. The DSST consists of 133 digits and requires the subject to substitute each digit with a simple symbol in a 90-second period. The number of correct symbols within the allowed time (eg, 90 sec) is measured. It takes approximately 5 minutes to complete and score the DSST.
Time Frame: Baseline to endpoint (week 8)
Population: as for outcome 1
Measure: Mean (Full Range); unit: number of correct symbols within 90 sec
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
number of correct symbols within 90 sec
  Baseline | 48.24 [30 to 65]
  Endpoint (week 8): number analyzed (Participants) | 22
  Endpoint (week 8) | 55.55 [30 to 73]
Statistical Analysis 1: Comparison: Vortioxetine; Test type: Other; p = 0.012, Paired t-test

3. Primary Outcome: BNA Scores Amplitudes
Description: Brain Network Analytics (BNA) is a tool intended for the post-hoc statistical analysis of the human EEG, utilizing both resting-state EEG and event-related potentials (ERP) waveforms. The BNA algorithm compares a patient's ERP amplitudes and latencies to those of a large group of healthy, age-matched subjects in order to visualize and quantify changes in specific brain functions. The BNA algorithm was used to detect subjects' P200 and P300 ERP components from EEG data recorded during the AOB and VGNG tasks. BNA scores represent these ERP components in terms of amplitude (in microvolts) and latency (in milliseconds).
Time Frame: Baseline to Endpoint (8 weeks)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
microvolts
  AOB P200 amplitude Baseline | 4.04 (2.60)
  AOB P200 amplitude Endpoint (8 weeks) | 3.96 (2.31)
  AOB P3a amplitude Baseline | 9.43 (5.00)
  AOB P3a amplitude Endpoint (8 weeks) | 7.13 (4.10)
  AOB P3b amplitude Baseline | 6.48 (3.69)
  AOB P3b amplitude Endpoint (8 weeks) | 6.75 (4.30)
  VGNG P200 amplitude Baseline | 3.40 (1.37)
  VGNG P200 amplitude Endpoint (8 weeks) | 3.66 (1.53)
  VGNG P3a amplitude Baseline | 3.33 (1.60)
  VGNG P3a amplitude Endpoint (8 weeks) | 3.55 (1.77)
Statistical Analysis 1: Comparison: Vortioxetine; Correlation between MADRS and AOB P200 (amplitude) baseline scores; Test type: Other; p = 0.610, Pearson's correlation; Pearson's R = 0.125
Statistical Analysis 2: Comparison: Vortioxetine; Correlation between MADRS and AOB P3a (amplitude) baseline scores; Test type: Other; p = 0.288, Pearson's correlation; Pearson's R = -0.294
Statistical Analysis 3: Comparison: Vortioxetine; Correlation between MADRS and AOB P3b (amplitude) baseline scores; Test type: Other; p = 0.134, Pearson's correlation; Pearson's R = -0.405
Statistical Analysis 4: Comparison: Vortioxetine; Correlation between MADRS and VGNG P200 (amplitude) baseline scores; Test type: Other; p = 0.083, Pearson's correlation; Pearson's R = -0.397
Statistical Analysis 5: Comparison: Vortioxetine; Correlation between MADRS and VGNG P3a (amplitude) baseline scores; Test type: Other; p = 0.034, Pearson's correlation; Pearson's R = -0.476
Statistical Analysis 6: Comparison: Vortioxetine; Correlation between DSST and AOB P200 baseline scores; Test type: Other; p = 0.031, Pearson's correlation; Pearson's R = -0.509
Statistical Analysis 7: Comparison: Vortioxetine; Correlation between DSST and AOB P3a (amplitude) baseline scores; Test type: Other; p = 0.500, Pearson's correlation; Pearson's R = -0.197
Statistical Analysis 8: Comparison: Vortioxetine; Correlation between DSST and AOB P3b baseline scores; Test type: Other; p = 0.185, Pearson's correlation; Pearson's R = 0.376
Statistical Analysis 9: Comparison: Vortioxetine; Correlation between DSST and VGNG P200 baseline scores; Test type: Other; p = 0.659, Pearson's correlation; Pearson's R = -0.108
Statistical Analysis 10: Comparison: Vortioxetine; Correlation between DSST and VGNG P3a baseline scores; Test type: Other; p = 0.611, Pearson's correlation; Pearson's R = 0.125
Statistical Analysis 11: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and MADRS (baseline to endpoint percent change); Test type: Other; p = 0.671, Pearson's correlation; Pearson's R = -0.111
Statistical Analysis 12: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and MADRS (baseline to endpoint percent change); Test type: Other; p = 0.931, Pearson's correlation; Pearson's R = -0.026
Statistical Analysis 13: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and MADRS (baseline to endpoint percent change); Test type: Other; p = 0.155, Pearson's correlation; Pearson's R = 0.516
Statistical Analysis 14: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and MADRS (baseline to endpoint percent change); Test type: Other; p = 0.297, Pearson's correlation; Pearson's R = 0.268
Statistical Analysis 15: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and MADRS (baseline to endpoint percent change); Test type: Other; p = 0.494, Pearson's correlation; Pearson's R = 0.184
Statistical Analysis 16: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and DSST (baseline to endpoint percent change); Test type: Other; p = 0.811, Pearson's correlation; Pearson's R = -0.065
Statistical Analysis 17: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and DSST (baseline to endpoint percent change); Test type: Other; p = 0.877, Pearson's correlation; Pearson's R = -0.048
Statistical Analysis 18: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and DSST (baseline to endpoint percent change); Test type: Other; p = 0.557, Pearson's correlation; Pearson's R = -0.246
Statistical Analysis 19: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and DSST (baseline to endpoint percent change); Test type: Other; p = 0.500, Pearson's correlation; Pearson's R = 0.182
Statistical Analysis 20: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and DSST (baseline to endpoint percent change); Test type: Other; p = 0.297, Pearson's correlation; Pearson's R = 0.288
Statistical Analysis 21: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P200 amplitudes at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other — Differences in BNA scores between MDD and healthy subjects were analyzed for baseline visits using an ANCOVA model with group as a factor, and age as a covariate; p = 0.575, ANCOVA; F statistic = 0.318
Statistical Analysis 22: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P200 amplitudes at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.541, ANCOVA; F statistic = 0.378
Statistical Analysis 23: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3a amplitudes at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.912, ANCOVA; F = 0.012
Statistical Analysis 24: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3a amplitudes at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.214, ANCOVA; F statistic = 1.586
Statistical Analysis 25: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3b amplitudes at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.504, ANCOVA; F statistic = 0.453
Statistical Analysis 26: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3b amplitudes at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.546, ANCOVA; F statistic = 0.37
Statistical Analysis 27: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P200 amplitudes at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.895, ANCOVA; F statistic = 0.017
Statistical Analysis 28: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P200 amplitudes at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.673, ANCOVA; F statistic = 0.179
Statistical Analysis 29: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P3a amplitudes at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.27, ANCOVA; F statistic = 1.241
Statistical Analysis 30: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P3a amplitudes at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.837, ANCOVA; F statistic = 0.042

4. Primary Outcome: BNA Scores Latencies
Description: as for outcome 3
Time Frame: Baseline to Endpoint (8 weeks)
Population: These correlation analyses were done only on participants in the vortioxetine arm and did not include the group of healthy controls
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
milliseconds
  AOB P200 latency Baseline | 177.37 (12.66)
  AOB P200 latency Endpoint (8 weeks) | 177.90 (14.12)
  AOB P3a latency Baseline | 308.47 (50.93)
  AOB P3a latency Endpoint (8 weeks) | 281.38 (40.63)
  AOB P3b latency Baseline | 370.07 (55.87)
  AOB P3b latency Endpoint (8 weeks) | 367.27 (37.59)
  VGNG P200 latency Baseline | 170.35 (14.05)
  VGNG P200 latency Endpoint (8 weeks) | 172.11 (16.35)
  VGNG P3a latency Baseline | 433.75 (24.91)
  VGNG P3a latency Endpoint (8 weeks) | 431.44 (32.36)
Statistical Analysis 1: Comparison: Vortioxetine; Correlation between DSST and AOB P200 (Latency) baseline scores; Test type: Other; p = 0.143, Pearson's correlation; Pearson's R = 0.359
Statistical Analysis 2: Comparison: Vortioxetine; Correlation between DSST and AOB P3b (latency) baseline scores; Test type: Other; p = 0.500, Pearson's correlation; Pearson's R = -0.197
Statistical Analysis 3: Comparison: Vortioxetine; Correlation between DSST and AOB P3b (latency) baseline scores; Test type: Other; p = 0.337, Pearson's correlation; Pearson's R = 0.277
Statistical Analysis 4: Comparison: Vortioxetine; Correlation between DSST and VGNG P200 (latency) baseline scores; Test type: Other; p = 0.832, Pearson's correlation; Pearson's R = 0.052
Statistical Analysis 5: Comparison: Vortioxetine; Correlation between DSST and VGNG P3a (latency) baseline scores; Test type: Other; p = 0.68, Pearson's correlation; Pearson's R = 0.103
Statistical Analysis 6: Comparison: Vortioxetine; Correlation between DSST and AOB P200 (Latency) baseline to endpoint percentage change; Test type: Other; p = 0.777, Pearson's correlation; Pearson's R = -0.074
Statistical Analysis 7: Comparison: Vortioxetine; Correlation between DSST and AOB P3a (Latency) baseline to endpoint percentage change; Test type: Other; p = 0.834, Pearson's correlation; Pearson's R = 0.061
Statistical Analysis 8: Comparison: Vortioxetine; Correlation between DSST and AOB P3b (Latency) baseline to endpoint percentage change; Test type: Other; p = 0.988, Pearson's correlation; Pearson's R = -0.006
Statistical Analysis 9: Comparison: Vortioxetine; Correlation between DSST and VGNG P200 (Latency) baseline to endpoint percentage change; Test type: Other; p = 0.788, Pearson's correlation; Pearson's R = 0.073
Statistical Analysis 10: Comparison: Vortioxetine; Correlation between DSST and VGNG P3a (Latency) baseline to endpoint percentage change; Test type: Other; p = 0.168, Pearson's correlation; Pearson's R = 0.375
Statistical Analysis 11: Comparison: Vortioxetine; Correlation between MADRS and AOB P200 (Latency) baseline scores; Test type: Other; p = 0.108, Pearson's correlation; Pearson's R = -0.392
Statistical Analysis 12: Comparison: Vortioxetine; Correlation between MADRS and AOB P3a (Latency) baseline scores; Test type: Other; p = 0.124, Pearson's correlation; Pearson's R = 0.415
Statistical Analysis 13: Comparison: Vortioxetine; Correlation between MADRS and AOB P3b (Latency) baseline scores; Test type: Other; p = 0.185, Pearson's correlation; Pearson's R = 0.362
Statistical Analysis 14: Comparison: Vortioxetine; Correlation between MADRS and VGNG P200 (Latency) baseline scores; Test type: Other; p = 0.923, Pearson's correlation; Pearson's R = -0.023
Statistical Analysis 15: Comparison: Vortioxetine; Correlation between MADRS and VGNG P3a (Latency) baseline scores; Test type: Other; p = 0.77, Pearson's correlation; Pearson's R = 0.071
Statistical Analysis 16: Comparison: Vortioxetine; Correlation between MADRS and AOB P200 (Latency) baseline to endpoint percent change; Test type: Other; p = 0.712, Pearson's correlation; Pearson's R = 0.097
Statistical Analysis 17: Comparison: Vortioxetine; Correlation between MADRS and AOB P3a (Latency) baseline to endpoint percent change; Test type: Other; p = 0.845, Pearson's correlation; Pearson's R = -0.058
Statistical Analysis 18: Comparison: Vortioxetine; Correlation between MADRS and AOB P3b (Latency) baseline to endpoint percent change; Test type: Other; p = 0.616, Pearson's correlation; Pearson's R = 0.194
Statistical Analysis 19: Comparison: Vortioxetine; Correlation between MADRS and VGNG P200 (Latency) baseline to endpoint percent change; Test type: Other; p = 0.323, Pearson's correlation; Pearson's R = 0.255
Statistical Analysis 20: Comparison: Vortioxetine; Correlation between MADRS and VGNG P3a (Latency) baseline to endpoint percent change; Test type: Other; p = 0.473, Pearson's correlation; Pearson's R = -0.193
Statistical Analysis 21: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P200 latencies at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.031, ANCOVA; F statistic = 4.909
Statistical Analysis 22: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P200 latencies at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.281, ANCOVA; F statistic = 1.189
Statistical Analysis 23: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3a latencies at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.966, ANCOVA; F statistic = 0.001
Statistical Analysis 24: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3a latencies at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.048, ANCOVA; F statistic = 4.121
Statistical Analysis 25: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3b latencies at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.005, ANCOVA; F statistic = 8.573
Statistical Analysis 26: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' AOB P3b latencies at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.101, ANCOVA; F statistic = 2.823
Statistical Analysis 27: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P200 latencies at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.373, ANCOVA; F statistic = 0.806
Statistical Analysis 28: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P200 latencies at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.183, ANCOVA; F statistic = 1.822
Statistical Analysis 29: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P3a latencies at baseline. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.475, ANCOVA; F statistic = 0.516
Statistical Analysis 30: Comparison: Vortioxetine; A comparison between vortioxetine arm patients' and healthy controls' VGNG P3a latencies at Endpoint. The healthy control group subjects have been previously documented in NCT02418208 (Clinical trials of the Rockies, Inc. Denver, Colorado, US and Clinical Research Center of Nevada Las Vegas, Nevada, US ) and in NCT02875496 (The Villages Health, The Villages, Florida, US); Test type: Other; p = 0.645, ANCOVA; F statistic = 0.214

5. Secondary Outcome: Changes in Hamilton Depression Rating Scale (HDRS) 17 From Baseline to 8 Week Endpoint
Description: The HDRS is a clinician-rated used to rate the patient's depressive state. The 17 question version of the scale rates depressive state based on feelings of depression, guilt, suicidality, anxiety, agitation, somatic symptoms, level of insight, patterns of insomnia, loss of interest in work and other activities, weight loss, and hypochondriasis. Additionally, the 28 question version rates depersonalization, paranoia, obsessions/compulsions, hypersomnia, appetite increase, and psychomotor slowing. The total score is obtained by summing the score of each item, 0-4 (symptom is absent, mild, moderate, or severe) or 0-2 (absent, slight or trivial, clearly present). Scores can range from 0 to 54 for the 17 question version and 0 to 83 for the 28 question version. Scores between 0 and 6 do not indicate the presence of depression, scores between 7 and 17 indicate mild depression, scores between 18 and 24 indicate moderate depression, and scores over 24 indicate severe depression.
Time Frame: Baseline to endpoint (week 8)
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
score on a scale
  Baseline | 23.76 [15 to 33]
  Endpoint (week 8): number analyzed (Participants) | 22
  Endpoint (week 8) | 11.59 [3 to 23]
Statistical Analysis 1: Comparison: Vortioxetine; Test type: Other; p < 0.001, Paired t-test

6. Secondary Outcome: Changes in Hamilton Depression Rating Scale (HDRS) 28 From Baseline to 8 Week Endpoint
Description: as for outcome 5
Time Frame: Baseline to endpoint (week 8)
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Vortioxetine: Open-label vortioxetine: 5-20 mg
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
score on a scale
  Baseline | 28.44 [19 to 40]
  Endpoint (week 8): number analyzed (Participants) | 22
  Endpoint (week 8) | 14.77 [3 to 26]
Statistical Analysis 1: Comparison: Vortioxetine; Test type: Other; p < 0.001, Paired t-test

7. Secondary Outcome: Changes in Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-16-SR) From Baseline to 8 Week Endpoint
Description: The QIDS-16-SR is a 16-item self-rated assessment of the severity of depressive symptoms. The assessments can be used to screen for depression, although they have been used predominantly as measures of symptom severity. The nine domains comprise 1) sad mood; 2) concentration; 3) self-criticism; 4) suicidal ideation; 5) interest; 6) energy/fatigue; 7) sleep disturbance (initial, middle, and late insomnia or hypersomnia); 8) decrease or increase in appetite or weight; and 9) psychomotor agitation or retardation. The total score ranges from 0 to 27 with higher scores equating to more severe symptomatology. The seven day period prior to assessment is the usual time frame for assessing symptom severity.
Time Frame: Baseline to endpoint (week 8)
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
score on a scale
  Baseline | 16.24 [9 to 21]
  Endpoint (week 8): number analyzed (Participants) | 22
  Endpoint (week 8) | 7.91 [0 to 18]
Statistical Analysis 1: Comparison: Vortioxetine; Test type: Other; p < 0.001, Paired t-test

8. Secondary Outcome: Changes in Clinical Global Impression Scale (CGI-S) From Baseline to 8 Week Endpoint
Description: The CGI-S assesses the clinician's impression of the subject's current mental illness state (considering their total clinical experience with this particular population) via 7 point scale (ranging from 1-7) with higher scores equating to more symptoms. For example, a score of 1 = normal, not at all ill and a score of 7 = severely ill.
Time Frame: Baseline to endpoint (week 8)
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
score on a scale
  Baseline | 4.88 [4 to 6]
  Endpoint (week 8): number analyzed (Participants) | 22
  Endpoint (week 8) | 2.64 [1 to 5]
Statistical Analysis 1: Comparison: Vortioxetine; Test type: Other; p < 0.001, Paired t-test

9. Secondary Outcome: Correlations Between BNA Amplitude Scores and Clinical, Cognitive, and Functionality Assessments Using Baseline Scores
Description: Pearson correlation was used to examine the associations between baseline BNA amplitude scores and outcomes including measures of MDD symptoms, cognitive function and functionality.
Time Frame: Baseline to Endpoint (8 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
microvolts
  AOB P200 amplitude Baseline | 4.04 (2.60)
  AOB P200 amplitude Endpoint (8 weeks) | 3.96 (2.31)
  AOB P3a amplitude Baseline | 9.43 (5.00)
  AOB P3a amplitude Endpoint (8 weeks) | 7.13 (4.10)
  AOB P3b amplitude Baseline | 6.48 (3.69)
  AOB P3b amplitude Endpoint (8 weeks) | 6.75 (4.30)
  VGNG P200 amplitude Baseline | 3.40 (1.37)
  VGNG P200 amplitude Endpoint (8 weeks) | 3.66 (1.53)
  VGNG P3a amplitude Baseline | 3.33 (1.60)
  VGNG P3a amplitude Endpoint (8 weeks) | 3.55 (1.77)
Statistical Analysis 1: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and HDRS-28 baseline scores; Test type: Other; p = 0.859, Pearson's correlation; Pearson's R = -0.044
Statistical Analysis 2: Comparison: Vortioxetine; AOB P3a (amplitude); Test type: Other; p = 0.451, Pearson's correlation; Pearson's R = -0.211
Statistical Analysis 3: Comparison: Vortioxetine; AOB P3b (amplitude); Test type: Other; p = 0.957, Pearson's correlation; Pearson's R = 0.015
Statistical Analysis 4: Comparison: Vortioxetine; VGNG P200 (amplitude); Test type: Other; p = 0.166, Pearson's correlation; Pearson's R = -0.322
Statistical Analysis 5: Comparison: Vortioxetine; VGNG P3a (amplitude); Test type: Other; p = 0.105, Pearson's correlation; Pearson's R = -0.374
Statistical Analysis 6: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and HDRS-28 baseline to endpoint percent change; Test type: Other; p = 0.601, Pearson's correlation; Pearson's R = -0.137
Statistical Analysis 7: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and HDRS-28 baseline to endpoint percent change; Test type: Other; p = 0.421, Pearson's correlation; Pearson's R = -0.234
Statistical Analysis 8: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and HDRS-28 baseline to endpoint percent change; Test type: Other; p = 0.316, Pearson's correlation; Pearson's R = 0.378
Statistical Analysis 9: Comparison: Vortioxetine; Test type: Other; p = 0.478, Pearson's correlation; Pearson's R = 0.185
Statistical Analysis 10: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and HDRS-28 baseline to endpoint percent change; Test type: Other; p = 0.969, Pearson's correlation; Pearson's R = 0.011
Statistical Analysis 11: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and HDRS-17 baseline scores; Test type: Other; p = 0.943, Pearson's correlation; Pearson's R = -0.018
Statistical Analysis 12: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and HDRS-17 baseline scores; Test type: Other; p = 0.795, Pearson's correlation; Pearson's R = -0.074
Statistical Analysis 13: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and HDRS-17 baseline scores; Test type: Other; p = 0.969, Pearson's correlation; Pearson's R = -0.011
Statistical Analysis 14: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and HDRS-17 baseline scores; Test type: Other; p = 0.406, Pearson's correlation; Pearson's R = -0.197
Statistical Analysis 15: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and HDRS-17 baseline scores; Test type: Other; p = 0.185, Pearson's correlation; Pearson's R = -0.309
Statistical Analysis 16: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.454, Pearson's correlation; Pearson's R = -0.195
Statistical Analysis 17: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.579, Pearson's correlation; Pearson's R = -0.162
Statistical Analysis 18: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.549, Pearson's correlation; Pearson's R = 0.232
Statistical Analysis 19: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.518, Pearson's correlation; Pearson's R = 0.169
Statistical Analysis 20: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.922, Pearson's correlation; Pearson's R = 0.027
Statistical Analysis 21: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and QIDS-SR baseline scores; Test type: Other; p = 0.796, Pearson's correlation; Pearson's R = -0.064
Statistical Analysis 22: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and QIDS-SR baseline scores; Test type: Other; p = 0.054, Pearson's correlation; Pearson's R = -0.506
Statistical Analysis 23: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and QIDS-SR baseline scores; Test type: Other; p = 0.995, Pearson's correlation; Pearson's R = 0.002
Statistical Analysis 24: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and QIDS-SR baseline scores; Test type: Other; p = 0.668, Pearson's correlation; Pearson's R = 0.102
Statistical Analysis 25: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and QIDS-SR baseline scores; Test type: Other; p = 0.875, Pearson's correlation; Pearson's R = 0.037
Statistical Analysis 26: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.852, Pearson's correlation; Pearson's R = -0.049
Statistical Analysis 27: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.234, Pearson's correlation; Pearson's R = -0.340
Statistical Analysis 28: Comparison: Vortioxetine; Test type: Other; p = 0.056, Pearson's correlation; Pearson's R = 0.655
Statistical Analysis 29: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.248, Pearson's correlation; Pearson's R = 0.297
Statistical Analysis 30: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.507, Pearson's correlation; Pearson's R = 0.179
Statistical Analysis 31: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and PDQ baseline scores; Test type: Other; p = 0.841, Pearson's correlation; Pearson's R = 0.049
Statistical Analysis 32: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and PDQ baseline scores; Test type: Other; p = 0.508, Pearson's correlation; Pearson's R = -0.185
Statistical Analysis 33: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and PDQ baseline scores; Test type: Other; p = 0.916, Pearson's correlation; Pearson's R = -0.030
Statistical Analysis 34: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and PDQ baseline scores; Test type: Other; p = 0.147, Pearson's correlation; Pearson's R = -0.345
Statistical Analysis 35: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and PDQ baseline scores; Test type: Other; p = 0.225, Pearson's correlation; Pearson's R = -0.284
Statistical Analysis 36: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.868, Pearson's correlation; Pearson's R = -0.044
Statistical Analysis 37: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.537, Pearson's correlation; Pearson's R = -0.180
Statistical Analysis 38: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.195, Pearson's correlation; Pearson's R = 0.476
Statistical Analysis 39: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.015, Pearson's correlation; Pearson's R = 0.594
Statistical Analysis 40: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.972, Pearson's correlation; Pearson's R = -0.009
Statistical Analysis 41: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and MGH-CPFQ baseline scores; Test type: Other; p = 0.785, Pearson's correlation; Pearson's R = 0.067
Statistical Analysis 42: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and MGH-CPFQ baseline scores; Test type: Other; p = 0.646, Pearson's correlation; Pearson's R = -0.129
Statistical Analysis 43: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and MGH-CPFQ baseline scores; Test type: Other; p = 0.182, Pearson's correlation; Pearson's R = 0.364
Statistical Analysis 44: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and MGH-CPFQ baseline scores; Test type: Other; p = 0.069, Pearson's correlation; Pearson's R = -0.414
Statistical Analysis 45: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and MGH-CPFQ baseline scores; Test type: Other; p = 0.068, Pearson's correlation; Pearson's R = -0.416
Statistical Analysis 46: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.929, Pearson's correlation; Pearson's R = -0.023
Statistical Analysis 47: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.802, Pearson's correlation; Pearson's R = -0.074
Statistical Analysis 48: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.153, Pearson's correlation; Pearson's R = 0.518
Statistical Analysis 49: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.298, Pearson's correlation; Pearson's R = 0.268
Statistical Analysis 50: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.996, Pearson's correlation; Pearson's R = -0.001
Statistical Analysis 51: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and WLQ baseline scores; Test type: Other; p = 0.531, Pearson's correlation; Pearson's R = 0.242
Statistical Analysis 52: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and WLQ baseline scores; Test type: Other; p = 0.210, Pearson's correlation; Pearson's R = -0.598
Statistical Analysis 53: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and WLQ baseline scores; Test type: Other; p = 0.899, Pearson's correlation; Pearson's R = 0.054
Statistical Analysis 54: Comparison: Vortioxetine; Test type: Other; p = 0.087, Pearson's correlation; Pearson's R = 0.568
Statistical Analysis 55: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and WLQ baseline scores; Test type: Other; p = 0.087, Pearson's correlation; Pearson's R = 0.568
Statistical Analysis 56: Comparison: Vortioxetine; Correlation between AOB P200 (amplitude) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.550, Pearson's correlation; Pearson's R = 0.231
Statistical Analysis 57: Comparison: Vortioxetine; Correlation between AOB P3a (amplitude) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.766, Pearson's correlation; Pearson's R = 0.158
Statistical Analysis 58: Comparison: Vortioxetine; Correlation between AOB P3b (amplitude) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.498, Pearson's correlation; Pearson's R = -0.406
Statistical Analysis 59: Comparison: Vortioxetine; Correlation between VGNG P200 (amplitude) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.599, Pearson's correlation; Pearson's R = 0.221
Statistical Analysis 60: Comparison: Vortioxetine; Correlation between VGNG P3a (amplitude) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.064, Pearson's correlation; Pearson's R = 0.679

10. Secondary Outcome: Correlations Between BNA Latency Scores and Clinical, Cognitive, and Functionality Assessments Using Baseline Scores
Description: Pearson correlation was used to examine the associations between baseline BNA latency scores and outcomes including measures of MDD symptoms, cognitive function and functionality.
Time Frame: Baseline to Endpoint (8 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Vortioxetine
Number analyzed (Participants) | 25
milliseconds
  AOB P200 latency Baseline | 177.37 (12.66)
  AOB P200 latency Endpoint (8 weeks) | 177.90 (14.12)
  AOB P3a latency Baseline | 308.47 (50.93)
  AOB P3a latency Endpoint (8 weeks) | 281.38 (40.63)
  AOB P3b latency Baseline | 370.07 (55.87)
  AOB P3b latency Endpoint (8 weeks) | 367.27 (37.59)
  VGNG P200 latency Baseline | 170.35 (14.05)
  VGNG P200 latency Endpoint (8 weeks) | 172.11 (16.35)
  VGNG P3a latency Baseline | 433.75 (24.91)
  VGNG P3a latency Endpoint (8 weeks) | 431.44 (32.36)
Statistical Analysis 1: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and HDRS-28 baseline scores; Test type: Other; p = 0.881, Pearson's correlation; Pearson's R = -0.038
Statistical Analysis 2: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and HDRS-28 baseline scores; Test type: Other; p = 0.279, Pearson's correlation; Pearson's R = 0.299
Statistical Analysis 3: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and HDRS-28 baseline scores; Test type: Other; p = 0.039, Pearson's correlation; Pearson's R = 0.538
Statistical Analysis 4: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and HDRS-28 baseline scores; Test type: Other; p = 0.940, Pearson's correlation; Pearson's R = -0.018
Statistical Analysis 5: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and HDRS-28 baseline scores; Test type: Other; p = 0.65, Pearson's correlation; Pearson's R = 0.107
Statistical Analysis 6: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and HDRS-28 baseline to endpoint percentage change; Test type: Other; p = 0.340, Pearson's correlation; Pearson's R = 0.247
Statistical Analysis 7: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and HDRS-28 baseline to endpoint percentage change; Test type: Other; p = 0.819, Pearson's correlation; Pearson's R = 0.067
Statistical Analysis 8: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and HDRS-28 baseline to endpoint percentage change; Test type: Other; p = 0.400, Pearson's correlation; Pearson's R = 0.321
Statistical Analysis 9: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and HDRS-28 baseline to endpoint percentage change; Test type: Other; p = 0.278, Pearson's correlation; Pearson's R = 0.279
Statistical Analysis 10: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and HDRS-28 baseline to endpoint percentage change; Test type: Other; p = 0.614, Pearson's correlation; Pearson's R = -0.136
Statistical Analysis 11: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and HDRS-17 baseline scores; Test type: Other; p = 0.999, Pearson's correlation; Pearson's R = 0.000
Statistical Analysis 12: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and HDRS-17 baseline scores; Test type: Other; p = 0.491, Pearson's correlation; Pearson's R = 0.193
Statistical Analysis 13: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and HDRS-17 baseline scores; Test type: Other; p = 0.028, Pearson's correlation; Pearson's R = 0.567
Statistical Analysis 14: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and HDRS-17 baseline scores; Test type: Other; p = 0.900, Pearson's correlation; Pearson's R = -0.030
Statistical Analysis 15: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and HDRS-17 baseline scores; Test type: Other; p = 0.55, Pearson's correlation; Pearson's R = 0.141
Statistical Analysis 16: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.373, Pearson's correlation; Pearson's R = 0.231
Statistical Analysis 17: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.949, Pearson's correlation; Pearson's R = 0.019
Statistical Analysis 18: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.754, Pearson's correlation; Pearson's R = 0.122
Statistical Analysis 19: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.499, 0.176; Pearson's R = 0.176
Statistical Analysis 20: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and HDRS-17 baseline to endpoint percent change; Test type: Other; p = 0.549, Pearson's correlation; Pearson's R = -0.162
Statistical Analysis 21: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and QIDS-SR baseline scores; Test type: Other; p = 0.617, Pearson's correlation; Pearson's R = -0.126
Statistical Analysis 22: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and QIDS-SR baseline scores; Test type: Other; p = 0.722, Pearson's correlation; Pearson's R = 0.100
Statistical Analysis 23: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and QIDS-SR baseline scores; Test type: Other; p = 0.371, Pearson's correlation; Pearson's R = 0.249
Statistical Analysis 24: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and QIDS-SR baseline scores; Test type: Other; p = 0.764, Pearson's correlation; Pearson's R = -0.072
Statistical Analysis 25: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and QIDS-SR baseline scores; Test type: Other; p = 0.34, Pearson's correlation; Pearson's R = -0.225
Statistical Analysis 26: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.570, Pearson's correlation; Pearson's R = 0.148
Statistical Analysis 27: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.434, Pearson's correlation; Pearson's R = 0.228
Statistical Analysis 28: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.569, Pearson's correlation; Pearson's R = 0.220
Statistical Analysis 29: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.005, Pearson's correlation; Pearson's R = 0.645
Statistical Analysis 30: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and QIDS-SR baseline to endpoint percent change; Test type: Other; p = 0.698, Pearson's correlation; Pearson's R = 0.105
Statistical Analysis 31: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and PDQ baseline scores; Test type: Other; p = 0.774, Pearson's correlation; Pearson's R = -0.073
Statistical Analysis 32: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and PDQ baseline score; Test type: Other; p = 0.024, Pearson's correlation; Pearson's R = 0.577
Statistical Analysis 33: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and PDQ baseline scores; Test type: Other; p = 0.603, Pearson's correlation; Pearson's R = 0.146
Statistical Analysis 34: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and PDQ baseline scores; Test type: Other; p = 0.326, Pearson's correlation; Pearson's R = -0.232
Statistical Analysis 35: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and PDQ baseline scores; Test type: Other; p = 0.68, Pearson's correlation; Pearson's R = 0.098
Statistical Analysis 36: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.774, Pearson's correlation; Pearson's R = -0.073
Statistical Analysis 37: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.024, Pearson's correlation; Pearson's R = 0.577
Statistical Analysis 38: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.603, Pearson's correlation; Pearson's R = 0.146
Statistical Analysis 39: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.326, Pearson's correlation; Pearson's R = -0.232
Statistical Analysis 40: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and PDQ baseline to endpoint percent change; Test type: Other; p = 0.68, Pearson's correlation; Pearson's R = 0.098
Statistical Analysis 41: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and MGH-CPFQ baseline scores; Test type: Other; p = 0.692, Pearson's correlation; Pearson's R = -0.100
Statistical Analysis 42: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and MGH-CPFQ baseline scores; Test type: Other; p = 0.059, Pearson's correlation; Pearson's R = 0.498
Statistical Analysis 43: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and MGH-CPFQ baseline scores; Test type: Other; p = 0.227, Pearson's correlation; Pearson's R = -0.332
Statistical Analysis 44: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and MGH-CPFQ baseline scores; Test type: Other; p = 0.600, Pearson's correlation; Pearson's R = -0.125
Statistical Analysis 45: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and MGH-CPFQ baseline scores; Test type: Other; p = 0.69, Pearson's correlation; Pearson's R = -0.096
Statistical Analysis 46: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.315, Pearson's correlation; Pearson's R = 0.259
Statistical Analysis 47: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.996, Pearson's correlation; Pearson's R = 0.002
Statistical Analysis 48: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.544, Pearson's correlation; Pearson's R = 0.234
Statistical Analysis 49: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.066, Pearson's correlation; Pearson's R = 0.455
Statistical Analysis 50: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and MGH-CPFQ baseline to endpoint percent change; Test type: Other; p = 0.293, Pearson's correlation; Pearson's R = -0.280
Statistical Analysis 51: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and WLQ baseline scores; Test type: Other; p = 0.013, Pearson's correlation; Pearson's R = 0.783
Statistical Analysis 52: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and WLQ baseline scores; Test type: Other; p = 0.799, Pearson's correlation; Pearson's R = 0.135
Statistical Analysis 53: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and WLQ baseline scores; Test type: Other; p = 0.201, Pearson's correlation; Pearson's R = 0.506
Statistical Analysis 54: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and WLQ baseline scores; Test type: Other; p = 0.586, Pearson's correlation; Pearson's R = -0.197
Statistical Analysis 55: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and WLQ baseline scores; Test type: Other; p = 0.95, Pearson's correlation; Pearson's R = -0.024
Statistical Analysis 56: Comparison: Vortioxetine; Correlation between AOB P200 (latency) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.920, Pearson's correlation; Pearson's R = 0.039
Statistical Analysis 57: Comparison: Vortioxetine; Correlation between AOB P3a (latency) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.831, Pearson's correlation; Pearson's R = 0.113
Statistical Analysis 58: Comparison: Vortioxetine; Correlation between AOB P3b (latency) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.230, Pearson's correlation; Pearson's R = 0.655
Statistical Analysis 59: Comparison: Vortioxetine; Correlation between VGNG P200 (latency) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.115, Pearson's correlation; Pearson's R = -0.602
Statistical Analysis 60: Comparison: Vortioxetine; Correlation between VGNG P3a (latency) and WLQ baseline to endpoint percent change; Test type: Other; p = 0.450, Pearson's correlation; Pearson's R = -0.313

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 9/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=25)
Nausea (Gastrointestinal disorders) | 9
Headache (General disorders) | 7
Upper respiratory infection (General disorders) | 6
Insomnia (General disorders) | 4
Somnolence (General disorders) | 3
Diarrhea (Gastrointestinal disorders) | 4
Esophageal reflux (General disorders) | 2
Sweating (General disorders) | 2
Dental/tooth pain (General disorders) | 2

LIMITATIONS AND CAVEATS:
Secondary outcomes #4 and #7, part c were not included in the results section for the following reasons: analysis became too complex based on low sample size; too many subgroups were needed. There were changes in BNA regardless of changes in symptoms and couldn't isolate meaningful or clinical useful data. In addition, several cognitive and functionality scores (i.e., CGI-I, TMT, UPSA, Stroop) were not collected at baseline and therefore not included in the "correlation with BNA" analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT02749721/Prot_SAP_000.pdf
  • Informed Consent Form: Consent version 08-29-16 IRB APPROVED (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT02749721/ICF_001.pdf
  • Informed Consent Form: onsent version 08-29-16 IRB APPROVED for 2017 (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT02749721/ICF_002.pdf
  • Informed Consent Form: consent version 04-09-18 IRB APPROVED (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT02749721/ICF_003.pdf